CLINICAL TRIAL: NCT01725308
Title: Phase II/III Study of FK949E: Placebo-controlled, Double-blind, Parallel-group Comparative Study and Open-label, Non-controlled Extension Study in Bipolar Disorder Patients With Major Depressive Episodes
Brief Title: A Study to Evaluate the Efficacy of FK949E in Bipolar Disorder Patients With Major Depressive Episodes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6949-CL-0021
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Bipolar Disorder
Keywords: FK949E; Major depressive episode; patients
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Participants who received placebo once daily at bedtime for 8 weeks in Treatment Period I and were evaluated against the transition criteria to transfer to Treatment Period II. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter. If transition criteria were met, participants went into Treatment Period II.
  Interventions: Drug: Placebo
- FK949E 150 mg (Experimental): After 2 days of up-titration, participants who received FK949E 150 mg once daily at bedtime for 8 weeks in Treatment Period I and were evaluated against the transition criteria to transfer to Treatment Period II. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter. If transition criteria were met, participants went into Treatment Period II.
  Interventions: Drug: FK949E
- FK949E 300 mg (Experimental): After 4 days of up-titration, participants who received FK949E 300 mg once daily at bedtime for 8 weeks in Treatment Period I and were evaluated against the transition criteria to transfer to Treatment Period II. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter. If transition criteria were met, participants went into Treatment Period II.
  Interventions: Drug: FK949E
- Placebo / FK949E (Experimental): Participants received placebo administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive placebo for 4 weeks, followed by a 1-week dose adjustment period, and a treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
  Interventions: Drug: FK949E; Drug: Placebo
- FK949E 150 mg / FK949E (Experimental): After 2 days of up-titration, participants received FK949E 150 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive FK949E 150 mg for 4 weeks followed by a 1-week dose-adjustment period and a treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
  Interventions: Drug: FK949E
- FK949E 300 mg / FK949E (Experimental): After 4 days of up-titration, participants received FK949E 300 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive FK949E 300 mg for 4 weeks followed by a 1-week dose-adjustment period and a treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — Taken by mouth (orally).
  Other Names: quetiapine
  Arms: FK949E 150 mg; FK949E 150 mg / FK949E; FK949E 300 mg; FK949E 300 mg / FK949E; Placebo / FK949E
Drug: Placebo — Taken by mouth (orally).
  Arms: Placebo; Placebo / FK949E

SUMMARY:
In period I, the treatment effect of FK949E was compared with that of placebo in a blind manner in bipolar disorder patients with major depressive episodes. In period II, the long-term safety and efficacy of FK949E was evaluated.

DETAILED DESCRIPTION:
This study consisted of two parts. In Treatment Period I, FK949E or placebo was administered orally in a blind manner to bipolar disorder patients with major depressive episodes, with the aim of evaluating the superiority of FK949E over placebo and the dose response of two doses of FK949E based on changes in Montgomery-Asberg Depression Rating Scale (MADRS) total score. In Treatment Period II, the long-term safety, efficacy and pharmacokinetics of open-label FK949E was evaluated in patients who completed Treatment Period I. An analysis was performed for data in Treatment Period I and another analysis was done for data in combined Treatment Periods I and II.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I or II disorder as specified in the Diagnostic and Statistical Manual of Mental Disorders Ver. 4 Text Revision (DSM-IV-TR,) with a major depressive episode
* The Hamilton Depression Rating Scale (HAM-D17) total score of 20 points or more and HAM-D17 depressed mood score of 2 points or more
* Able to participate in the study with understanding of and compliance with subject requirements during the study in the investigator's or subinvestigator's opinion

Exclusion Criteria:

* Concurrent or previous history of DSM-IV-TR Axis I disorders, except bipolar disorder, within the last 6 months before informed consent
* Concurrence of DSM-IV-TR Axis II disorder that is considered to greatly affect patient's current mental status
* The Young Mania Rating Scale (YMRS) total score of 13 points or more
* Nine or more mood episodes within the last 12 months before informed consent
* Lack of response to at least 6-week treatment with at least 2 antidepressants for the current major depressive episode in the investigator's or subinvestigator's opinion
* History of abuse or dependence of alcohol or substances other than caffeine and nicotine
* Treatment with a depot antipsychotic within the last 42 days before primary registration
* Unable to stop taking mood stabilizers (lithium carbonate and/or sodium valproate), lamotrigine, antipsychotics, or antidepressants from 7 days before secondary registration
* Unable to stop taking antiepileptics (except lamotrigine and sodium valproate), antianxiety agents, hypnotics, sedatives, psychostimulants, antiparkinsonian agents, cerebral ameliorators, antidementia agents, or anorectics, except those specified as conditionally-allowed concomitant drugs, after primary registration
* Electroconvulsive therapy within the last 76 days before primary registration
* The current major depressive episode persisting for more than 12 months or less than 4 weeks before informed consent
* A possible need of psychotherapy during the study period (unless the therapy has been commenced at least 76 days before primary registration and been maintained on a fixed level at fixed frequency)
* Documented or suspected conditions such as renal failure, hepatic failure, serious cardiac disease, hepatitis B, hepatitis C, or acquired immunodeficiency syndrome (AIDS) (or to be a carrier of hepatitis B, hepatitis C, or AIDS)
* Concurrence of malignancy or history of cured malignancy within 5 years
* Concurrence of uncontrolled hypertension (defined as a systolic blood pressure of 180 mmHg or more, or a diastolic blood pressure of 110 mmHg or more at primary registration) or unstable angina that may worsen with the study or may affect the study results based on the clinical judgment of the investigator or sub-investigator
* Concurrence of hypotension (defined as a systolic blood pressure of less than 100 mmHg at primary registration) or orthostatic hypotension
* History of transient, idiopathic orthostatic hypotension, with or without pre-syncope symptoms or syncope, or a current condition susceptible to transient hypotension, such as dehydration and decreased blood volume
* Concurrent or previous history of cerebrovascular disease or transient ischemic attack (TIA)
* Abnormal laboratory or electrocardiographic findings considered clinically significant in the investigator's or subinvestigator's opinion (in reference to grade 3 of the Adverse Drug Reactions Severity Grading Criteria [Notification No. 80 of the Safety Division, Pharmaceutical Affairs Bureau, Ministry of Health and Welfare dated 29 June 1992])
* Participation in another clinical study or post-marketing study within the last 12 weeks before informed consent
* History of quetiapine therapy during the current major depressive episode
* Pregnant or lactating women

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 431 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (98):
- Japan (98):
  - Site JP00030, Aichi
  - Site JP00031, Aichi
  - Site JP00052, Aichi
  - Site JP00055, Aichi
  - Site JP00072, Aichi
  - Site JP00092, Aichi
  - Site JP00003, Akita
  - Site JP00008, Chiba
  - Site JP00009, Chiba
  - Site JP00002, Fukuoka
  - Site JP00037, Fukuoka
  - Site JP00038, Fukuoka
  - Site JP00039, Fukuoka
  - Site JP00040, Fukuoka
  - Site JP00041, Fukuoka
  - Site JP00058, Fukuoka
  - Site JP00082, Fukuoka
  - Site JP00083, Fukuoka
  - Site JP00091, Fukuoka
  - Site JP00094, Fukuoka
  - Site JP00095, Fukuoka
  - Site JP00096, Fukuoka
  - Site JP00097, Fukuoka
  - Site JP00098, Fukuoka
  - Site JP00004, Fukushima
  - Site JP00028, Gifu
  - Site JP00006, Gunma
  - Site JP00007, Gunma
  - Site JP00035, Hiroshima
  - Site JP00056, Hiroshima
  - Site JP00067, Hiroshima
  - Site JP00001, Hokkaido
  - Site JP00059, Hokkaido
  - Site JP00061, Hokkaido
  - Site JP00062, Hokkaido
  - Site JP00068, Hokkaido
  - Site JP00069, Hokkaido
  - Site JP00073, Hokkaido
  - Site JP00074, Hokkaido
  - Site JP00076, Hokkaido
  - Site JP00005, Ibaraki
  - Site JP00049, Kagawa
  - Site JP00021, Kanagawa
  - Site JP00022, Kanagawa
  - Site JP00023, Kanagawa
  - Site JP00024, Kanagawa
  - Site JP00025, Kanagawa
  - Site JP00042, Kumamoto
  - Site JP00050, Kumamoto
  - Site JP00032, Kyoto
  - Site JP00084, Kyoto
  - Site JP00077, Miyagi
  - Site JP00027, Nagano
  - Site JP00075, Nara
  - Site JP00054, Okayama
  - Site JP00079, Okayama
  - Site JP00043, Okinawa
  - Site JP00046, Okinawa
  - Site JP00033, Osaka
  - Site JP00034, Osaka
  - Site JP00047, Osaka
  - Site JP00063, Osaka
  - Site JP00053, Ōita
  - Site JP00029, Shizuoka
  - Site JP00036, Tokushima
  - Site JP00010, Tokyo
  - Site JP00011, Tokyo
  - Site JP00012, Tokyo
  - Site JP00013, Tokyo
  - Site JP00014, Tokyo
  - Site JP00015, Tokyo
  - Site JP00016, Tokyo
  - Site JP00017, Tokyo
  - Site JP00018, Tokyo
  - Site JP00019, Tokyo
  - Site JP00020, Tokyo
  - Site JP00045, Tokyo
  - Site JP00048, Tokyo
  - Site JP00051, Tokyo
  - Site JP00057, Tokyo
  - Site JP00060, Tokyo
  - Site JP00064, Tokyo
  - Site JP00065, Tokyo
  - Site JP00066, Tokyo
  - Site JP00070, Tokyo
  - Site JP00071, Tokyo
  - Site JP00078, Tokyo
  - Site JP00081, Tokyo
  - Site JP00085, Tokyo
  - Site JP00086, Tokyo
  - Site JP00087, Tokyo
  - Site JP00088, Tokyo
  - Site JP00089, Tokyo
  - Site JP00090, Tokyo
  - Site JP00093, Tokyo
  - Site JP00099, Tokyo
  - Site JP00044, Tottori
  - Site JP00026, Toyama

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fukushi R, Nomura Y, Katashima M, Komatsu K, Sato Y, Takada A. Approach to Evaluating QT Prolongation of Quetiapine Fumarate in Late Stage of Clinical Development Using Concentration-QTc Modeling and Simulation in Japanese Patients With Bipolar Disorder. Clin Ther. 2020 Aug;42(8):1483-1493.e1. doi: 10.1016/j.clinthera.2020.06.002. Epub 2020 Aug 11. PMID 32792252
- [Derived] Fukushi R, Nomura Y, Katashima M, Komatsu K, Sato Y, Takada A. Population Pharmacokinetics Analysis of Quetiapine Extended-release Formulation in Japanese Patients with Bipolar Depression. Clin Ther. 2020 Jun;42(6):1067-1076.e2. doi: 10.1016/j.clinthera.2020.04.006. Epub 2020 Jun 6. PMID 32518042
- [Derived] Kanba S, Murasaki M, Koyama T, Takeuchi M, Shimizu Y, Arita E, Kuroishi K, Takeuchi M, Kamei S. Long-term mood/antidepressant effects of quetiapine extended-release formulation: an open-label, non-controlled extension study in Japanese patients with bipolar depression. BMC Psychiatry. 2019 Jun 26;19(1):198. doi: 10.1186/s12888-019-2181-9. PMID 31242884
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese patients with bipolar I or bipolar II as specified in Diagnostic and Statistical Manual of Mental Disorders Ver. 4 Text Revision (DSM-IV-TR) whose most recent episode was diagnosed as a major depressive episode using the Mini-International Neuropsychiatric Interview (MINI) were recruited for this study.
Pre-assignment Details: Assignment of participants to the FK949E 150 mg group was discontinued with implementation of Version 3.0 of the protocol.
Period: Treatment Period I
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Started | 178 | 74 | 179
Treated | 177 | 74 | 179
Completed | 134 | 60 | 138
Not Completed | 44 | 14 | 41
Not completed — Did Not Receive Drug | 1 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 21
Not completed — Insufficient Response | 7 | 0 | 5
Not completed — Worsening of the Target Disease | 8 | 0 | 2
Not completed — Changes in the Episodes | 3 | 0 | 2
Not completed — Withdrawal of Consent | 12 | 7 | 5
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Protocol Deviations | 3 | 1 | 1
Not completed — Miscellaneous | 2 | 0 | 3
Period: Treatment Period II
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Started | 134 | 60 | 138
Treated | 120 | 53 | 130
Completed | 79 | 31 | 74
Not Completed | 55 | 29 | 64
Not completed — Did Not Meet Transition Criteria | 0 | 3 | 4
Not completed — Did Not Receive Drug | 4 | 0 | 0
Not completed — Adverse Event | 13 | 8 | 20
Not completed — Insufficient Response | 2 | 4 | 6
Not completed — Worsening of the Target Disease | 1 | 4 | 2
Not completed — Changes in the Episodes | 1 | 0 | 5
Not completed — Withdrawal of Consent | 28 | 2 | 16
Not completed — Lost to Follow-up | 1 | 5 | 3
Not completed — Protocol Deviations | 0 | 0 | 1
Not completed — Miscellaneous | 5 | 3 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), which included participants who received at least one dose of study drug and had measurements taken for at least one efficacy endpoint after start of drug treatment in Treatment Period I.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg | Total
Number analyzed (Participants) | 177 | 74 | 179 | 430
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (11.0) | 39.2 (10.2) | 38.1 (11.2) | 38.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 37 | 93 | 231
  Male | 76 | 37 | 86 | 199
Total Montgomery-Åsberg Depression Rating Scale (MADRS) score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
  units on a scale | 30.8 (6.4) | 30.2 (6.8) | 30.9 (6.9) | 30.7 (6.7)
Total Hamilton Depression Rating Scale (HAM-D17) Score [Mean (Standard Deviation); unit: units on a scale] — The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52, where a higher score indicates a greater depressive state.
  units on a scale | 23.1 (2.8) | 23.3 (3.4) | 23.0 (3.0) | 23.1 (3.0)
Number of Participants wirth MADRS Remission [Count of Participants; unit: Participants] — MADRS remission was defined as MADRS total score of 12 or less. The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
  Participants | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment Period I in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
Time Frame: Baseline and Week 8
Population: FAS; Last observation carried forward (LOCF) imputation was used for end of Treatment Period I.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale | -10.1 (10.9) | -14.4 (11.4) | -12.6 (11.4)
Statistical Analysis 1: Comparison: Placebo vs FK949E 300 mg; An analysis of covariance (ANCOVA) using a model where the total MADRS score at baseline is a covariate and the treatment group and bipolar disorder diagnosis (Type I/ II) are fixed effects; Test type: Superiority or Other; p = 0.034, ANCOVA; Least squares mean difference = -2.4, 95% CI 2-sided [-4.7 to -0.2]

2. Secondary Outcome: Change From Baseline in MADRS Total Score (Treatment Period I)
Description: as for outcome 1
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | -3.5 (5.4) | -6.4 (8.1) | -5.1 (6.8)
  Week 2 | -5.1 (7.0) | -10.0 (8.9) | -8.3 (8.6)
  Week 3 | -7.1 (8.8) | -11.6 (9.9) | -9.9 (9.3)
  Week 4 | -8.5 (9.1) | -12.5 (10.8) | -11.8 (9.5)
  Week 6 | -9.2 (10.1) | -14.5 (11.0) | -12.2 (10.9)
  Week 8 | -10.1 (10.9) | -14.4 (11.4) | -12.6 (11.4)

3. Secondary Outcome: Change From Baseline in MADRS Total Score (Combined Treatment Period I and II)
Description: The MADRS is a10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: Baseline (Week 0 for FK949E 150 mg/FK949E & FK949E 300 mg/FK949E and Week 12 for Placebo/FK949E) and Weeks 1, 2, 3, 4, 6, 8, 10, 12 13, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: FAS for combined Treatment Period I and II, which included participants who received at least one dose of FK949E and had measurements taken for at least one efficacy endpoint after the start of FK949E treatment, and with available data at each time point. LOCF imputation method was used at end of combined treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FK949E 300 mg / FK949E: After 4 days of up-titration, participants received FK949E 300 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive FK949E 300 mg for 4 weeks followed by a 1-week dose-adjustment period and treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | -6.4 (8.1) | -5.1 (6.8)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | -10.0 (8.9) | -8.5 (8.7)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | -12.0 (10.1) | -10.6 (9.3)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | -13.1 (11.0) | -13.2 (9.2)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | -15.6 (11.2) | -13.8 (10.8)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | -15.8 (11.5) | -14.8 (10.9)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | -16.3 (11.6) | -15.9 (10.9)
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | -16.4 (12.1) | -16.0 (10.3)
  Week 13: number analyzed (Participants) | 119 | 51 | 120
  Week 13 | -1.6 (5.8) | -18.1 (10.4) | -13.3 (10.1)
  Week 14: number analyzed (Participants) | 113 | 50 | 118
  Week 14 | -3.1 (7.0) | -17.0 (10.7) | -16.4 (10.7)
  Week 16: number analyzed (Participants) | 108 | 48 | 117
  Week 16 | -4.3 (7.7) | -17.1 (10.3) | -17.2 (10.2)
  Week 18: number analyzed (Participants) | 106 | 48 | 115
  Week 18 | -6.8 (8.0) | -17.3 (11.5) | -19.0 (9.8)
  Week 20: number analyzed (Participants) | 101 | 47 | 115
  Week 20 | -6.8 (8.3) | -18.7 (10.6) | -18.2 (9.9)
  Week 24: number analyzed (Participants) | 100 | 42 | 111
  Week 24 | -7.1 (8.5) | -21.4 (10.5) | -18.4 (10.2)
  Week 28: number analyzed (Participants) | 95 | 38 | 105
  Week 28 | -7.0 (8.6) | -22.9 (8.5) | -19.4 (10.4)
  Week 32: number analyzed (Participants) | 88 | 36 | 98
  Week 32 | -6.6 (10.2) | -22.3 (9.6) | -19.4 (10.3)
  Week 36: number analyzed (Participants) | 84 | 35 | 92
  Week 36 | -7.5 (9.4) | -23.1 (10.4) | -19.4 (10.5)
  Week 40: number analyzed (Participants) | 82 | 33 | 88
  Week 40 | -8.2 (9.8) | -23.3 (9.7) | -19.8 (10.4)
  Week 44: number analyzed (Participants) | 80 | 33 | 83
  Week 44 | -8.1 (10.0) | -23.4 (10.2) | -20.7 (9.7)
  Week 48: number analyzed (Participants) | 80 | 32 | 76
  Week 48 | -7.6 (10.0) | -24.1 (10.2) | -20.9 (10.7)
  Week 52: number analyzed (Participants) | 78 | 32 | 74
  Week 52 | -7.8 (10.7) | -24.4 (10.1) | -22.1 (9.3)
  End of combined treatment period | -6.6 (10.4) | -16.0 (13.3) | -15.2 (12.2)

4. Secondary Outcome: Number of Participants With MADRS Response (Treatment Period I)
Description: A MADRS response was defined as a decrease in MADRS total score of 50% or more from baseline. The MADRS is a10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
Participants
  Week 1 | 4 | 6 | 15
  Week 2 | 13 | 17 | 41
  Week 3 | 36 | 25 | 52
  Week 4 | 47 | 28 | 62
  Week 6 | 54 | 34 | 70
  Week 8 | 63 | 32 | 79

5. Secondary Outcome: Number of Participants With MADRS Response (Combined Treatment Period I and II)
Description: A MADRS response was defined as a decrease in MADRS total score of 50% or more from baseline. The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: Baseline (Week 0 for FK949E 150 mg/FK949E & FK949E 300 mg/FK949E and Week 12 for Placebo/FK949E) and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: FAS (for combined Treatment Period I and II) participants with available data at each time point; LOCF imputation method was used at end of combined treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 6 | 15
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 16 | 37
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | 23 | 49
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 25 | 58
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | 30 | 66
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | 27 | 73
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | 28 | 71
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | 22 | 68
  Week 13: number analyzed (Participants) | 113 | 51 | 120
  Week 13 | 8 | 32 | 65
  Week 14: number analyzed (Participants) | 107 | 50 | 118
  Week 14 | 26 | 30 | 66
  Week 16: number analyzed (Participants) | 102 | 48 | 117
  Week 16 | 31 | 26 | 67
  Week 18: number analyzed (Participants) | 100 | 48 | 115
  Week 18 | 48 | 30 | 78
  Week 20: number analyzed (Participants) | 95 | 47 | 115
  Week 20 | 47 | 30 | 73
  Week 24: number analyzed (Participants) | 94 | 42 | 111
  Week 24 | 48 | 31 | 74
  Week 28: number analyzed (Participants) | 89 | 38 | 105
  Week 28 | 48 | 34 | 71
  Week 32: number analyzed (Participants) | 83 | 36 | 98
  Week 32 | 43 | 31 | 65
  Week 36: number analyzed (Participants) | 79 | 35 | 92
  Week 36 | 43 | 30 | 61
  Week 40: number analyzed (Participants) | 77 | 33 | 88
  Week 40 | 47 | 28 | 62
  Week 44: number analyzed (Participants) | 75 | 33 | 83
  Week 44 | 42 | 28 | 61
  Week 48: number analyzed (Participants) | 75 | 32 | 76
  Week 48 | 38 | 29 | 57
  Week 52: number analyzed (Participants) | 73 | 32 | 74
  Week 52 | 41 | 27 | 57
  End of combined treatment period: number analyzed (Participants) | 114 | 74 | 179
  End of combined treatment period | 57 | 42 | 89

6. Secondary Outcome: Number of Participants With MADRS Remission (Treatment Period I)
Description: MADRS remission was defined as MADRS total score of 12 or less. The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
Participants
  Week 1 | 4 | 4 | 12
  Week 2 | 9 | 12 | 28
  Week 3 | 26 | 21 | 39
  Week 4 | 31 | 21 | 49
  Week 6 | 39 | 27 | 60
  Week 8 | 47 | 28 | 68

7. Secondary Outcome: Number of Participants With MADRS Remission (Combined Treatment Period I and II)
Description: MADRS remission was defined as MADRS total score of 12 or less. The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-10.
Time Frame: Weeks 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 4 | 12
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 11 | 25
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | 20 | 36
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 19 | 45
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | 24 | 56
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | 25 | 61
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | 24 | 61
  Week 12: number analyzed (Participants) | 119 | 49 | 120
  Week 12 | 41 | 20 | 58
  Week 13: number analyzed (Participants) | 120 | 51 | 120
  Week 13 | 48 | 24 | 58
  Week 14: number analyzed (Participants) | 114 | 50 | 118
  Week 14 | 51 | 24 | 60
  Week 16: number analyzed (Participants) | 109 | 48 | 117
  Week 16 | 52 | 20 | 60
  Week 18: number analyzed (Participants) | 107 | 48 | 115
  Week 18 | 69 | 23 | 68
  Week 20: number analyzed (Participants) | 102 | 47 | 115
  Week 20 | 64 | 24 | 64
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 67 | 28 | 65
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 62 | 28 | 64
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 55 | 28 | 58
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 56 | 27 | 53
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 60 | 26 | 55
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 54 | 24 | 54
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 55 | 24 | 51
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 54 | 26 | 51
  End of combined treatment period | 75 | 38 | 82

8. Secondary Outcome: Change From Baseline in Hamilton Depression Rating Scale (HAM-D17) Total Score (Treatment Period I)
Description: The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52, where a higher score indicates a greater depressive state.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | -3.4 (4.2) | -5.9 (5.1) | -4.5 (4.9)
  Week 2 | -5.1 (5.4) | -8.7 (5.8) | -7.0 (6.0)
  Week 3 | -6.6 (6.5) | -10.0 (6.2) | -7.9 (6.2)
  Week 4 | -7.3 (6.7) | -10.9 (6.6) | -9.2 (6.4)
  Week 6 | -7.7 (7.3) | -11.9 (7.1) | -9.6 (7.0)
  Week 8 | -8.4 (7.6) | -11.9 (7.4) | -10.1 (7.6)
Statistical Analysis 1: Comparison: Placebo vs FK949E 300 mg; At End of Treatment Period I/Week 8: An analysis of covariance (ANCOVA) using a model where the total HAM-D17 score at baseline is a covariate and the treatment group and bipolar disorder diagnosis (Type I/II) are fixed effects; Test type: Superiority or Other; p = 0.033, ANCOVA; Least squares mean difference = -1.7, 95% CI 2-sided [-3.3 to -0.1]

9. Secondary Outcome: Change From Baseline in HAM-D17 (Combined Treatment Period I and II)
Description: The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52, where a higher score indicates a greater depressive state. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: Baseline (Week 0 for FK949E 150 mg/FK949E & FK949E 300 mg/FK949E and Week 12 for Placebo/FK949E) and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 28, 36, 40, 44, 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | -5.9 (5.1) | -4.5 (4.9)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | -8.8 (5.8) | -7.1 (5.8)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | -10.3 (6.0) | -8.4 (6.1)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | -11.4 (6.5) | -9.9 (6.3)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | -12.7 (7.0) | -10.7 (6.8)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | -13.0 (7.1) | -11.6 (7.2)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | -13.1 (7.8) | -12.4 (7.2)
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | -13.7 (7.5) | -12.6 (6.5)
  Week 14: number analyzed (Participants) | 113 | 50 | 118
  Week 14 | -1.9 (4.7) | -13.9 (7.5) | -12.8 (7.1)
  Week 16: number analyzed (Participants) | 108 | 48 | 117
  Week 16 | -2.9 (5.2) | -13.7 (7.1) | -13.4 (6.9)
  Week 20: number analyzed (Participants) | 101 | 47 | 115
  Week 20 | -4.2 (6.0) | -14.6 (7.3) | -13.8 (6.6)
  Week 28: number analyzed (Participants) | 95 | 38 | 105
  Week 28 | -4.8 (6.0) | -16.7 (6.4) | -14.3 (7.0)
  Week 36: number analyzed (Participants) | 84 | 35 | 92
  Week 36 | -4.9 (6.4) | -17.1 (6.9) | -14.6 (6.8)
  Week 44: number analyzed (Participants) | 80 | 33 | 83
  Week 44 | -5.7 (7.0) | -17.0 (7.6) | -15.1 (6.9)
  Week 52: number analyzed (Participants) | 78 | 32 | 74
  Week 52 | -5.6 (7.1) | -17.8 (7.9) | -16.2 (6.7)
  End of combined treatment period | -4.6 (6.6) | -12.9 (8.7) | -11.6 (8.3)

10. Secondary Outcome: Number of Participants With HAM-D17 Response (Treatment Period I)
Description: A HAM-D17 response was defined as a decrease in HAM-D17 total score of 50% or more from baseline. The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52, where a higher score indicates a greater depressive state.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
Participants
  Week 1 | 10 | 7 | 14
  Week 2 | 29 | 22 | 42
  Week 3 | 41 | 30 | 52
  Week 4 | 54 | 35 | 64
  Week 6 | 63 | 44 | 66
  Week 8 | 68 | 41 | 78

11. Secondary Outcome: Number of Participants With HAM-D17 Response (Combined Treatment Period I and II)
Description: A HAM-D17 response was defined as a decrease in HAM-D17 total score of 50% or more from baseline. The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52, where a higher score indicates a greater depressive state. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: Baseline (Week 0 for FK949E 150 mg/FK949E & FK949E 300 mg/FK949E and Week 12 for Placebo/FK949E) and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 28, 36, 44, 52
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 7 | 14
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 22 | 39
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | 27 | 50
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 32 | 61
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | 39 | 63
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | 35 | 73
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | 35 | 77
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | 32 | 77
  Week 14: number analyzed (Participants) | 109 | 50 | 118
  Week 14 | 20 | 35 | 78
  Week 16: number analyzed (Participants) | 104 | 48 | 117
  Week 16 | 30 | 30 | 80
  Week 20: number analyzed (Participants) | 97 | 47 | 115
  Week 20 | 40 | 32 | 75
  Week 28: number analyzed (Participants) | 91 | 38 | 105
  Week 28 | 44 | 32 | 73
  Week 36: number analyzed (Participants) | 80 | 35 | 92
  Week 36 | 36 | 29 | 61
  Week 44: number analyzed (Participants) | 76 | 33 | 83
  Week 44 | 41 | 25 | 61
  Week 52: number analyzed (Participants) | 74 | 32 | 74
  Week 52 | 40 | 25 | 58
  End of combined treatment period: number analyzed (Participants) | 116 | 74 | 179
  End of combined treatment period | 53 | 43 | 95

12. Secondary Outcome: Change From Baseline in Clinical Global Impression-Bipolar Disorder-Severity (CGI-BP-S): Mania (Treatment Period I)
Description: The CGI-BP-S is a scale which assesses a participant's severity of their overall bipolar illness, depression, and mania as assessed by the clinician using a scale from 1 (not ill) to 7 (very severely ill).
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | -0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2)
  Week 2 | -0.0 (0.2) | -0.0 (0.2) | 0.0 (0.2)
  Week 3 | 0.0 (0.2) | -0.0 (0.2) | 0.0 (0.2)
  Week 4 | 0.0 (0.2) | -0.0 (0.4) | 0.0 (0.2)
  Week 6 | 0.0 (0.3) | -0.1 (0.2) | 0.0 (0.3)
  Week 8 | 0.0 (0.3) | -0.1 (0.4) | 0.0 (0.2)

13. Secondary Outcome: Change From Baseline in CGI-BP-S: Mania (Combined Treatment Period I and II)
Description: The CGI-BP-S is a scale which assesses a participant's severity of their overall bipolar illness, depression, and mania as assessed by the clinician using a scale from 1 (not ill) to 7 (very severely ill). Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: Baseline (Week 0 for FK949E 150 mg/FK949E & FK949E 300 mg/FK949E and Week 12 for Placebo/FK949E) and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 0.0 (0.2) | 0.0 (0.2)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 0.0 (0.2) | -0.0 (0.2)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | -0.0 (0.2) | 0.0 (0.1)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 0.0 (0.4) | 0.0 (0.1)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | -0.0 (0.2) | 0.0 (0.2)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | -0.0 (0.4) | -0.0 (0.2)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | -0.0 (0.3) | 0.0 (0.1)
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | 0.0 (0.1) | -0.0 (0.2)
  Week 14: number analyzed (Participants) | 113 | 50 | 118
  Week 14 | -0.0 (0.3) | -0.1 (0.2) | -0.0 (0.2)
  Week 16: number analyzed (Participants) | 108 | 48 | 117
  Week 16 | -0.0 (0.3) | -0.1 (0.2) | -0.0 (0.2)
  Week 18: number analyzed (Participants) | 106 | 48 | 115
  Week 18 | -0.0 (0.3) | -0.1 (0.2) | -0.0 (0.2)
  Week 20: number analyzed (Participants) | 101 | 47 | 115
  Week 20 | -0.0 (0.3) | -0.1 (0.2) | -0.0 (0.2)
  Week 24: number analyzed (Participants) | 100 | 42 | 111
  Week 24 | -0.0 (0.2) | -0.0 (0.3) | 0.0 (0.2)
  Week 28: number analyzed (Participants) | 95 | 38 | 105
  Week 28 | -0.0 (0.2) | -0.0 (0.3) | 0.0 (0.3)
  Week 32: number analyzed (Participants) | 88 | 36 | 98
  Week 32 | -0.0 (0.2) | 0.0 (0.3) | 0.0 (0.5)
  Week 36: number analyzed (Participants) | 84 | 35 | 92
  Week 36 | -0.0 (0.2) | -0.0 (0.3) | -0.0 (0.1)
  Week 40: number analyzed (Participants) | 82 | 33 | 88
  Week 40 | -0.0 (0.2) | 0.0 (0.3) | 0.0 (0.2)
  Week 44: number analyzed (Participants) | 80 | 33 | 83
  Week 44 | -0.0 (0.2) | -0.0 (0.2) | -0.0 (0.1)
  Week 48: number analyzed (Participants) | 80 | 32 | 76
  Week 48 | -0.0 (0.2) | -0.0 (0.2) | 0.0 (0.2)
  Week 52: number analyzed (Participants) | 78 | 32 | 74
  Week 52 | -0.0 (0.2) | -0.0 (0.2) | -0.0 (0.1)
  End of combined treatment period | -0.0 (0.3) | -0.1 (0.3) | 0.1 (0.5)

14. Secondary Outcome: Change From Baseline in CGI-BP-S: Depression (Treatment Period I)
Description: The CGI-BP-S is a scale which assesses a participant's severity of their overall bipolar illness, depression, and mania as assessed by the clinician with the scale from 1 (not ill) to 7 (very severely ill).
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | -0.3 (0.7) | -0.5 (0.8) | -0.4 (0.7)
  Week 2 | -0.5 (0.9) | -0.8 (1.0) | -0.7 (1.0)
  Week 3 | -0.7 (1.1) | -1.0 (1.1) | -0.9 (1.0)
  Week 4 | -0.8 (1.1) | -1.2 (1.2) | -1.1 (1.0)
  Week 6 | -0.9 (1.2) | -1.3 (1.2) | -1.1 (1.2)
  Week 8 | -1.0 (1.4) | -1.4 (1.3) | -1.2 (1.3)

15. Secondary Outcome: Change From Baseline in CGI-BP-S: Depression (Combined Treatment Period I and II)
Description: as for outcome 13
Time Frame: as for outcome 13
Population: FAS (for combined Treatment Period I and II) participants with available data at each time point; LOCF imputation was used at end of combined treatment period.
Measure: Mean (Standard Deviation); unit: units on a sale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a sale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | -0.5 (0.8) | -0.4 (0.7)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | -0.8 (1.1) | -0.7 (1.0)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | -1.0 (1.2) | -1.0 (1.0)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | -1.2 (1.2) | -1.2 (1.0)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | -1.4 (1.2) | -1.3 (1.2)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | -1.5 (1.3) | -1.5 (1.3)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | -1.5 (1.4) | -1.6 (1.3)
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | -1.5 (1.4) | -1.7 (1.2)
  Week 14: number analyzed (Participants) | 113 | 50 | 118
  Week 14 | -0.3 (0.7) | -1.5 (1.4) | -1.7 (1.3)
  Week 16: number analyzed (Participants) | 108 | 48 | 117
  Week 16 | -0.5 (0.8) | -1.7 (1.3) | -1.7 (1.3)
  Week 18: number analyzed (Participants) | 106 | 48 | 115
  Week 18 | -0.7 (0.9) | -1.7 (1.4) | -2.0 (1.3)
  Week 20: number analyzed (Participants) | 101 | 47 | 115
  Week 20 | -0.7 (1.0) | -1.8 (1.4) | -1.9 (1.3)
  Week 24: number analyzed (Participants) | 100 | 42 | 111
  Week 24 | -0.8 (1.1) | -2.1 (1.4) | -2.0 (1.3)
  Week 28: number analyzed (Participants) | 95 | 38 | 105
  Week 28 | -0.8 (1.2) | -2.4 (1.2) | -2.0 (1.3)
  Week 32: number analyzed (Participants) | 88 | 36 | 98
  Week 32 | -0.8 (1.3) | -2.4 (1.4) | -2.1 (1.2)
  Week 36: number analyzed (Participants) | 84 | 35 | 92
  Week 36 | -0.9 (1.2) | -2.6 (1.4) | -2.0 (1.2)
  Week 40: number analyzed (Participants) | 82 | 33 | 88
  Week 40 | -0.9 (1.3) | -2.5 (1.3) | -2.1 (1.3)
  Week 44: number analyzed (Participants) | 80 | 33 | 83
  Week 44 | -0.9 (1.3) | -2.3 (1.4) | -2.2 (1.1)
  Week 48: number analyzed (Participants) | 80 | 32 | 76
  Week 48 | -0.9 (1.3) | -2.5 (1.3) | -2.3 (1.3)
  Week 52: number analyzed (Participants) | 78 | 32 | 74
  Week 52 | -0.9 (1.4) | -2.7 (1.3) | -2.4 (1.2)
  End of combined treatment period | -0.8 (1.4) | -1.8 (1.6) | -1.6 (1.5)

16. Secondary Outcome: Change From Baseline in CGI-BP-S: Overall Bipolar Illness (Treatment Period I)
Description: as for outcome 14
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | -0.3 (0.7) | -0.4 (0.8) | -0.4 (0.7)
  Week 2 | -0.5 (0.9) | -0.7 (1.0) | -0.7 (0.9)
  Week 3 | -0.7 (1.0) | -0.9 (1.1) | -0.9 (1.0)
  Week 4 | -0.8 (1.1) | -1.1 (1.1) | -1.1 (1.0)
  Week 6 | -0.8 (1.2) | -1.2 (1.2) | -1.1 (1.2)
  Week 8 | -1.0 (1.3) | -1.4 (1.3) | -1.2 (1.3)

17. Secondary Outcome: Change From Baseline in CGI-BP-S: Overall Bipolar Illness (Combined Treatment Period I and II)
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | -0.4 (0.8) | -0.4 (0.7)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | -0.7 (1.0) | -0.7 (1.0)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | -0.9 (1.1) | -1.0 (1.0)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | -1.1 (1.2) | -1.2 (1.0)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | -1.3 (1.2) | -1.3 (1.2)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | -1.4 (1.3) | -1.5 (1.3)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | -1.4 (1.4) | -1.6 (1.4)
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | -1.4 (1.5) | -1.7 (1.2)
  Week 14: number analyzed (Participants) | 113 | 50 | 118
  Week 14 | -0.3 (0.7) | -1.4 (1.4) | -1.6 (1.3)
  Week 16: number analyzed (Participants) | 108 | 48 | 117
  Week 16 | -0.5 (0.8) | -1.6 (1.3) | -1.7 (1.3)
  Week 18: number analyzed (Participants) | 106 | 48 | 115
  Week 18 | -0.7 (0.9) | -1.6 (1.4) | -1.9 (1.3)
  Week 20: number analyzed (Participants) | 101 | 47 | 115
  Week 20 | -0.8 (1.0) | -1.7 (1.4) | -1.9 (1.3)
  Week 24: number analyzed (Participants) | 100 | 42 | 111
  Week 24 | -0.8 (1.0) | -2.0 (1.4) | -1.9 (1.3)
  Week 28: number analyzed (Participants) | 95 | 38 | 105
  Week 28 | -0.9 (1.1) | -2.2 (1.3) | -1.9 (1.3)
  Week 32: number analyzed (Participants) | 88 | 36 | 98
  Week 32 | -0.8 (1.3) | -2.2 (1.4) | -2.0 (1.3)
  Week 36: number analyzed (Participants) | 84 | 35 | 92
  Week 36 | -0.9 (1.2) | -2.4 (1.5) | -2.0 (1.2)
  Week 40: number analyzed (Participants) | 82 | 33 | 88
  Week 40 | -1.0 (1.3) | -2.3 (1.3) | -2.1 (1.3)
  Week 44: number analyzed (Participants) | 80 | 33 | 83
  Week 44 | -1.0 (1.3) | -2.2 (1.5) | -2.2 (1.2)
  Week 48: number analyzed (Participants) | 80 | 32 | 76
  Week 48 | -0.9 (1.2) | -2.4 (1.5) | -2.3 (1.3)
  Week 52: number analyzed (Participants) | 78 | 32 | 74
  Week 52 | -1.0 (1.3) | -2.6 (1.4) | -2.4 (1.2)
  End of combined treatment period | -0.8 (1.3) | -1.7 (1.6) | -1.5 (1.5)

18. Secondary Outcome: Clinical Global Impression-Bipolar Disorder-Change (CGI-BP-C): Mania (Treatment Period I)
Description: The CGI-BP-C is a scale which assesses the degree of change or improvement from baseline for each of overall bipolar illness, depression and mania, by grading it using 8 grades, from 1 (very much improved) to 7 (very much worse) or 8 (not applicable). Grade 8 (not applicable) was regarded as a missing value for purposes of calculating the mean score.
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | 4.0 (0.3) | 4.0 (0.2) | 4.0 (0.1)
  Week 2 | 4.0 (0.2) | 4.0 (0.2) | 4.0 (0.3)
  Week 3 | 4.0 (0.2) | 4.0 (0.2) | 4.0 (0.2)
  Week 4 | 4.0 (0.3) | 4.0 (0.4) | 4.0 (0.2)
  Week 6 | 4.0 (0.3) | 3.9 (0.2) | 4.0 (0.3)
  Week 8 | 4.0 (0.3) | 3.9 (0.3) | 4.0 (0.2)

19. Secondary Outcome: CGI-BP-C: Mania (Combined Treatment Period I and II)
Description: The CGI-BP-C is a scale which assesses the degree of change or improvement from baseline for each of overall bipolar illness, depression and mania, by grading it using 8 grades, from 1 (very much improved) to 7 (very much worse) or 8 (not applicable). Grade 8 (not applicable) was regarded as a missing value for purposes of calculating the mean score. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-10.
Time Frame: Weeks 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52 (Placebo/FK949E only from week 12, FK949E 150 mg/FK949E & FK949E 300 mg/FK949E from week 1)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 4.0 (0.2) | 4.0 (0.1)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 4.0 (0.2) | 4.0 (0.3)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | 4.0 (0.2) | 4.0 (0.2)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 4.0 (0.3) | 4.0 (0.2)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | 4.0 (0.2) | 4.0 (0.3)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | 4.0 (0.3) | 4.0 (0.3)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | 4.0 (0.3) | 4.0 (0.2)
  Week 12: number analyzed (Participants) | 119 | 49 | 120
  Week 12 | 4.0 (0.4) | 4.0 (0.1) | 4.0 (0.2)
  Week 14: number analyzed (Participants) | 114 | 50 | 118
  Week 14 | 3.9 (0.5) | 4.0 (0.2) | 4.0 (0.2)
  Week 16: number analyzed (Participants) | 109 | 48 | 117
  Week 16 | 3.9 (0.5) | 4.0 (0.2) | 4.0 (0.2)
  Week 18: number analyzed (Participants) | 107 | 48 | 115
  Week 18 | 3.9 (0.5) | 4.0 (0.2) | 4.0 (0.1)
  Week 20: number analyzed (Participants) | 102 | 47 | 115
  Week 20 | 3.9 (0.5) | 4.0 (0.2) | 4.0 (0.2)
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 4.0 (0.5) | 4.0 (0.2) | 4.0 (0.2)
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 3.9 (0.4) | 4.0 (0.2) | 4.0 (0.2)
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 4.0 (0.4) | 4.0 (0.3) | 4.0 (0.3)
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 4.0 (0.3) | 4.0 (0.4) | 4.0 (0.1)
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 4.0 (0.3) | 4.0 (0.2) | 4.0 (0.2)
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 4.0 (0.4) | 4.0 (0.0) | 4.0 (0.1)
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 4.0 (0.4) | 4.0 (0.0) | 4.0 (0.2)
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 3.9 (0.4) | 4.0 (0.0) | 4.0 (0.1)
  End of combined treatment period | 4.0 (0.5) | 3.9 (0.3) | 4.1 (0.3)

20. Secondary Outcome: CGI-BP-C: Depression (Treatment Period I)
Description: as for outcome 18
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | 3.7 (0.8) | 3.5 (0.8) | 3.5 (0.8)
  Week 2 | 3.6 (1.0) | 3.1 (0.9) | 3.2 (1.0)
  Week 3 | 3.4 (1.2) | 2.9 (0.9) | 3.0 (1.1)
  Week 4 | 3.2 (1.3) | 2.8 (1.0) | 2.9 (1.2)
  Week 6 | 3.2 (1.3) | 2.7 (1.0) | 2.8 (1.2)
  Week 8 | 3.1 (1.4) | 2.6 (1.1) | 2.8 (1.2)

21. Secondary Outcome: CGI-BP-C: Depression (Combined Treatment Period I and II)
Description: as for outcome 19
Time Frame: as for outcome 19
Population: FAS (for combined Treatment Period I and II) participants with available data at each time point; LOCF imputtion was used at end of combined treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 3.5 (0.8) | 3.5 (0.8)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 3.1 (0.9) | 3.1 (1.0)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | 2.9 (0.9) | 2.9 (1.1)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 2.7 (1.0) | 2.7 (1.1)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | 2.6 (1.0) | 2.7 (1.1)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | 2.5 (1.1) | 2.5 (1.1)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | 2.5 (1.1) | 2.4 (1.1)
  Week 12: number analyzed (Participants) | 119 | 49 | 120
  Week 12 | 2.7 (1.2) | 2.6 (1.2) | 2.4 (1.0)
  Week 14: number analyzed (Participants) | 114 | 50 | 118
  Week 14 | 2.4 (1.2) | 2.6 (1.2) | 2.4 (1.1)
  Week 16: number analyzed (Participants) | 109 | 48 | 117
  Week 16 | 2.3 (1.2) | 2.4 (1.0) | 2.4 (1.1)
  Week 18: number analyzed (Participants) | 107 | 48 | 115
  Week 18 | 2.1 (1.2) | 2.5 (1.3) | 2.2 (1.1)
  Week 20: number analyzed (Participants) | 102 | 47 | 115
  Week 20 | 2.0 (1.0) | 2.3 (1.2) | 2.2 (1.2)
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 1.9 (0.9) | 2.1 (1.1) | 2.2 (1.1)
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 1.9 (0.9) | 1.9 (0.9) | 2.2 (1.2)
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 1.9 (1.0) | 2.0 (1.2) | 2.1 (1.1)
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 1.9 (1.0) | 1.8 (0.9) | 2.1 (1.1)
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 1.8 (1.0) | 1.8 (0.8) | 2.1 (1.1)
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 1.8 (0.9) | 2.0 (1.0) | 1.9 (0.9)
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 1.9 (1.0) | 1.9 (0.9) | 1.9 (1.1)
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 1.8 (1.0) | 1.7 (0.9) | 1.8 (1.0)
  End of combined period | 2.0 (1.2) | 2.5 (1.4) | 2.6 (1.4)

22. Secondary Outcome: CGI-BP-C: Overall Bipolar Illness (Treatment Period I)
Description: as for outcome 18
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: FAS; LOCF imputation method was used for all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 79
units on a scale
  Week 1 | 3.7 (0.8) | 3.5 (0.8) | 3.5 (0.8)
  Week 2 | 3.6 (1.0) | 3.1 (0.9) | 3.2 (1.0)
  Week 3 | 3.4 (1.2) | 2.9 (0.9) | 3.0 (1.1)
  Week 4 | 3.3 (1.3) | 2.8 (1.0) | 2.9 (1.2)
  Week 6 | 3.3 (1.4) | 2.7 (1.0) | 2.9 (1.2)
  Week 8 | 3.1 (1.5) | 2.6 (1.1) | 2.8 (1.2)

23. Secondary Outcome: CGI-BP-C: Overall Bipolar Illness (Combined Treatment Period I and II)
Description: as for outcome 19
Time Frame: as for outcome 19
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | 3.5 (0.8) | 3.5 (0.8)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | 3.1 (0.9) | 3.2 (1.0)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | 2.9 (0.9) | 2.9 (1.1)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | 2.7 (1.0) | 2.7 (1.1)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | 2.6 (1.1) | 2.7 (1.1)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | 2.5 (1.1) | 2.5 (1.1)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | 2.5 (1.1) | 2.4 (1.1)
  Week 12: number analyzed (Participants) | 119 | 49 | 120
  Week 12 | 2.7 (1.2) | 2.6 (1.2) | 2.4 (1.0)
  Week 14: number analyzed (Participants) | 114 | 50 | 118
  Week 14 | 2.4 (1.2) | 2.6 (1.2) | 2.4 (1.1)
  Week 16: number analyzed (Participants) | 109 | 48 | 117
  Week 16 | 2.3 (1.2) | 2.4 (1.0) | 2.4 (1.1)
  Week 18: number analyzed (Participants) | 107 | 48 | 115
  Week 18 | 2.1 (1.1) | 2.5 (1.3) | 2.2 (1.0)
  Week 20: number analyzed (Participants) | 102 | 47 | 115
  Week 20 | 2.0 (1.0) | 2.3 (1.2) | 2.3 (1.1)
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 1.9 (0.9) | 2.1 (1.1) | 2.2 (1.1)
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 1.9 (0.9) | 1.9 (0.9) | 2.2 (1.2)
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 2.0 (1.1) | 2.1 (1.2) | 2.2 (1.3)
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 1.9 (1.0) | 1.9 (1.1) | 2.1 (1.1)
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 1.8 (1.0) | 1.8 (0.8) | 2.1 (1.1)
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 1.8 (0.9) | 2.0 (1.0) | 1.9 (0.9)
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 1.9 (1.0) | 1.9 (1.0) | 2.0 (1.1)
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 1.8 (1.0) | 1.7 (0.9) | 1.8 (1.0)
  End of combined treatment period | 2.1 (1.2) | 2.5 (1.4) | 2.7 (1.5)

24. Secondary Outcome: Number of Participants With Adverse Events (Treatment Period I)
Description: An adverse event (AE) is defined as any undesirable or unintended sign (including abnormal laboratory test values), symptom, or disease occurring while the study drug was administered, regardless of whether or not there was a causal relationship with the study drug. A serious AE is defined as a an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important.
Time Frame: Up to 8 weeks
Population: Safety Analysis Set (SAF), which included participants who received at least one dose of study drug for Treatment Period I.
Measure: Number; unit: participants
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
participants
  Any AE | 81 | 55 | 149
  Drug-related AEs | 52 | 50 | 133
  Deaths | 1 | 0 | 0
  Serious AEs | 2 | 1 | 0
  Drug-related SAEs | 0 | 0 | 0
  AEs that caused study drug discontimuation | 16 | 6 | 27
  Drug-related AEs that caused study drug discont. | 11 | 5 | 23

25. Secondary Outcome: Number of Participants With Adverse Events (Combined Treatment Period I and II)
Description: An AE is defined as any undesirable or unintended sign (including abnormal laboratory test values), symptom, or disease occurring while the study drug was administered, regardless of whether or not there was a causal relationship with the study drug. A serious AE is defined as a an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. AEs reported are AEs that occurred after the start of the FK949E treatment for all groups.
Time Frame: Up to 54 weeks (Placebo / FK949E, from week 12 to week 52, for FK949E 150 mg / FK949E & FK949E 300 mg / FK949E groups, from week 0 to week 52)
Population: SAF for combined Treatment Periods I and II, which included participants who were treated with FK949E at least one time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Any AE | 110 | 63 | 171
  Drug-related AEs | 100 | 60 | 159
  Deaths | 0 | 0 | 0
  Serious AEs | 1 | 4 | 5
  Drug-related SAEs | 0 | 2 | 2
  AEs that caused study drug discontimuation | 15 | 15 | 51
  Drug-related AEs that caused study drug discont | 13 | 11 | 39

26. Secondary Outcome: Change From Baseline in Drug Induced Extra-Pyramidal Symptoms Scale (DIEPSS): Total Score (Treatment Period I)
Description: The DIEPSS is a scale used to evaluate drug-induced extrapyramidal symptoms. DIEPSS is composed of 8 individual symptom parameters and a global assessment of severity, each rated on a 5-point scale, with lower scores indicating as "normal." The DIEPSS total score ranges from 0 (none, normal) to 32 (severe), and excludes the global assessment of severity.
Time Frame: Baseline and Weeks 4, 8
Population: SAF participants with available data at each time point; LOCF was used for end of Treatment Period I.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment Period I: FK949E 300 mg: After 4 days of up-titration, participants who received FK949E 300 mg once daily at bedtime for 8 weeks in Treatment Period I and were evaluated against the transition criteria to transfer to Treatment Period II. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter. If transition criteria were met, participants went into Treatment Period II.
Arm/Group | Placebo | FK949E 150 mg | Treatment Period I: FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 4: number analyzed (Participants) | 160 | 68 | 159
  Week 4 | 0.0 (0.5) | 0.0 (0.7) | 0.2 (1.2)
  Week 8: number analyzed (Participants) | 136 | 60 | 140
  Week 8 | 0.1 (0.5) | 0.0 (0.7) | 0.1 (1.1)
  End of Treatment Period I: number analyzed (Participants) | 173 | 73 | 176
  End of Treatment Period I | 0.1 (0.6) | 0.0 (0.8) | 0.1 (1.1)

27. Secondary Outcome: Change From Baseline in DIEPSS: Total Score (Combined Treatment Period I and II)
Description: The DIEPSS is a scale used to evaluate drug-induced extrapyramidal symptoms. DIEPSS is composed of 8 individual symptom parameters and a global assessment of severity, each rated on a 5-point scale, with lower scores indicating as "normal." The DIEPSS total score ranges from 0 (none, normal) to 32 (severe), and excludes the global assessment of severity. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: Baseline (Week 0 for FK949E 150 mg/FK949E & FK949E 300 mg/FK949E and Week 12 for Placebo/FK949E) and Weeks 4, 8, 12, 16, 20, 28, 36, 44, 52
Population: SAF (for combined Treatment Period I and II) participants with available data at each time point; LOCF imputation was used at end of combined treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0.0 (0.7) | 0.2 (1.2)
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0.0 (0.7) | 0.1 (1.1)
  Week 12: number analyzed (Participants) | 0 | 51 | 123
  Week 12 |  | 0.1 (0.8) | 0.1 (1.0)
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0.2 (0.9) | 0.1 (0.7) | 0.1 (1.0)
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0.1 (0.8) | 0.1 (1.0) | 0.1 (1.0)
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0.1 (0.7) | -0.0 (0.6) | 0.0 (1.1)
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0.0 (0.7) | 0.0 (0.7) | -0.1 (0.8)
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0.0 (0.4) | -0.0 (0.6) | -0.1 (0.9)
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0.1 (0.5) | 0.0 (0.6) | -0.2 (1.0)
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 0.1 (0.7) | -0.0 (0.7) | 0.0 (1.0)

28. Secondary Outcome: Change From Baseline in DIEPSS: Parkinsonism (Treatment Period I)
Description: The DIEPSS is a scale used to evaluate drug-induced extrapyramidal symptoms. DIEPSS is composed of 8 individual symptom parameters and a global assessment of severity, each rated on a 5-point scale, with lower scores indicating as "normal." Parkinsonism is a total of the gait disturbance, bradykinesia, salivation, muscle rigidity, and tremor scores and ranges from 0 (none, normal) to 20 (severe).
Time Frame: Baseline and Weeks 4, 8
Population: SAF participants with available data at each time point; LOCF imputation method for end of Treatment Period I was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 4: number analyzed (Participants) | 160 | 68 | 159
  Week 4 | 0.0 (0.4) | -0.1 (0.5) | 0.0 (0.8)
  Week 8: number analyzed (Participants) | 136 | 60 | 140
  Week 8 | 0.0 (0.3) | -0.1 (0.5) | -0.1 (0.8)
  End of Treatment Period I: number analyzed (Participants) | 173 | 73 | 176
  End of Treatment Period I | 0.1 (0.4) | -0.1 (0.5) | -0.1 (0.7)

29. Secondary Outcome: Change From Baseline in DIEPSS: Parkinsonism (Combined Treatment Period I and II)
Description: The DIEPSS is a scale used to evaluate drug-induced extrapyramidal symptoms. DIEPSS is composed of 8 individual symptom parameters and a global assessment of severity, each rated on a 5-point scale, with lower scores indicating as "normal." Parkinsonism is a total of the gait disturbance, bradykinesia, salivation, muscle rigidity, and tremor scores and ranges from 0 (none, normal) to 20 (severe). Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: umits on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
umits on a scale
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | -0.1 (0.5) | 0.0 (0.8)
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | -0.1 (0.5) | -0.1 (0.8)
  Week 12: number analyzed (Participants) | 0 | 51 | 123
  Week 12 |  | 0.0 (0.7) | -0.1 (0.8)
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0.0 (0.7) | -0.0 (0.6) | -0.1 (0.8)
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0.0 (0.4) | -0.0 (0.7) | -0.1 (0.7)
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | -0.0 (0.3) | -0.1 (0.5) | -0.1 (0.8)
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | -0.1 (0.3) | -0.1 (0.5) | -0.1 (0.7)
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | -0.0 (0.2) | -0.1 (0.4) | -0.1 (0.8)
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | -0.0 (0.3) | -0.1 (0.4) | -0.2 (0.9)
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | -0.0 (0.4) | -0.1 (0.5) | -0.1 (0.7)

30. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) (Treatment Period I)
Description: The YMRS is a scale used to evaluate manic symptoms. The YMRS total score was the total assessment of assessed points for 11 items, ranges from 0 to 60 (each item is scored from either 0-4 or 0-8 by severity (0 = absent and 4/8 = displays mood/behavior to a greater degree). A lower score indicates "Absent" or "Normal."
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, 8
Population: SAF participants with available data at each time point; LOCF imputation method for end of Treatment Period I was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 177 | 74 | 179
units on a scale
  Week 1 | -0.1 (1.6) | -0.6 (1.8) | -0.6 (2.1)
  Week 2: number analyzed (Participants) | 165 | 72 | 162
  Week 2 | -0.2 (1.4) | -1.0 (1.5) | -0.7 (1.9)
  Week 3: number analyzed (Participants) | 158 | 67 | 157
  Week 3 | -0.1 (1.9) | -1.2 (1.7) | -0.7 (1.8)
  Week 4: number analyzed (Participants) | 146 | 66 | 150
  Week 4 | -0.4 (1.7) | -1.3 (2.0) | -0.9 (1.7)
  Week 6: number analyzed (Participants) | 144 | 62 | 147
  Week 6 | -0.3 (2.2) | -1.4 (2.1) | -0.8 (1.9)
  Week 8: number analyzed (Participants) | 135 | 59 | 138
  Week 8 | -0.4 (1.6) | -1.7 (2.3) | -0.9 (1.7)
  End of Treatment Period 1 | -0.2 (2.1) | -1.6 (2.3) | -0.8 (2.0)

31. Secondary Outcome: Change From Baseline in YMRS (Combined Treatment Period I and II)
Description: The YMRS is a scale used to evaluate manic symptoms. The YMRS total score was the total assessment of assessed points for 11 items, ranges from 0 to 60 (each item is scored from either 0-4 or 0-8 by severity (0 = absent and 4/8 = displays mood/behavior to a greater degree). A lower score indicates "Absent" or "Normal." Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-12.
Time Frame: as for outcome 5
Population: SAF (for combined Treatment Period I and II) participants with available data at each time point; LOCF imputation was used for value at end of combined treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
units on a scale
  Week 1: number analyzed (Participants) | 0 | 74 | 179
  Week 1 |  | -0.6 (1.8) | -0.6 (2.1)
  Week 2: number analyzed (Participants) | 0 | 72 | 162
  Week 2 |  | -1.0 (1.5) | -0.7 (1.9)
  Week 3: number analyzed (Participants) | 0 | 67 | 157
  Week 3 |  | -1.2 (1.7) | -0.7 (1.8)
  Week 4: number analyzed (Participants) | 0 | 66 | 150
  Week 4 |  | -1.3 (2.0) | -0.9 (1.7)
  Week 6: number analyzed (Participants) | 0 | 62 | 147
  Week 6 |  | -1.4 (2.1) | -0.8 (1.9)
  Week 8: number analyzed (Participants) | 0 | 59 | 138
  Week 8 |  | -1.7 (2.3) | -0.9 (1.7)
  Week 10: number analyzed (Participants) | 0 | 53 | 127
  Week 10 |  | -1.6 (2.1) | -0.8 (2.1)
  Week 12: number analyzed (Participants) | 0 | 49 | 120
  Week 12 |  | -1.2 (1.6) | -1.0 (1.7)
  Week 13: number analyzed (Participants) | 119 | 51 | 120
  Week 13 | -0.3 (1.5) | -1.3 (1.6) | -1.1 (1.5)
  Week 14: number analyzed (Participants) | 113 | 50 | 118
  Week 14 | -0.4 (1.7) | -1.6 (1.9) | -1.1 (1.4)
  Week 16: number analyzed (Participants) | 108 | 48 | 117
  Week 16 | -0.5 (1.8) | -1.3 (2.1) | -0.9 (1.6)
  Week 18: number analyzed (Participants) | 106 | 48 | 115
  Week 18 | -0.7 (1.9) | -1.6 (2.0) | -1.1 (1.9)
  Week 20: number analyzed (Participants) | 101 | 47 | 115
  Week 20 | -0.5 (1.8) | -1.5 (2.2) | -0.9 (1.8)
  Week 24: number analyzed (Participants) | 100 | 42 | 111
  Week 24 | -0.6 (1.9) | -1.4 (1.9) | -0.9 (2.1)
  Week 28: number analyzed (Participants) | 95 | 38 | 105
  Week 28 | -0.7 (1.9) | -1.6 (2.0) | -1.1 (2.0)
  Week 32: number analyzed (Participants) | 88 | 36 | 98
  Week 32 | -0.7 (1.6) | -1.4 (2.4) | -0.3 (5.1)
  Week 36: number analyzed (Participants) | 84 | 35 | 92
  Week 36 | -0.7 (1.9) | -1.3 (2.4) | -0.9 (1.8)
  Week 40: number analyzed (Participants) | 82 | 33 | 88
  Week 40 | -0.8 (1.8) | -1.6 (2.1) | -1.0 (2.0)
  Week 44: number analyzed (Participants) | 79 | 33 | 83
  Week 44 | -0.5 (2.0) | -1.7 (1.9) | -1.1 (1.8)
  Week 48: number analyzed (Participants) | 80 | 32 | 76
  Week 48 | -0.7 (1.7) | -1.9 (2.1) | -1.3 (1.5)
  Week 52: number analyzed (Participants) | 78 | 32 | 74
  Week 52 | -0.8 (1.8) | -1.9 (2.0) | -1.2 (1.6)
  End of combined treatment period: number analyzed (Participants) | 119 | 74 | 179
  End of combined treatment period | -0.5 (2.2) | -1.6 (2.0) | -0.4 (4.2)

32. Secondary Outcome: Number of Participants With an Affirmative Response to Columbia Suicide Severity Rating Scale (C-SSRS): Suicidal Ideation (Treatment Period I)
Description: The C-SSRS is a scale for assessing risk for suicidal behavior and suicide ideation and was administered by the clinician. Affirmative or negative responses were provided to 5 items for suicide ideation (1. Wish to be dead; 2. Suicidal thoughts; 3. Suicidal thoughts with a method (no specific plan or intent to act); 4. Suicidal intent (without a specific plan); 5. Suicidal intent with specific plan. If participants responded with a negative response for questions 1 and 2, the remaining questions are skipped. If question 2 was responded to with a positive response, the remaining questions need to be asked.
Time Frame: Weeks 4, 8
Population: SAF participants with available data at each time point; LOCF imputation method was used for end of Treatment Period I.
Measure: Number; unit: participants
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 173 | 73 | 176
participants
  Week 4: Wish to be dead: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Wish to be dead | 39 | 14 | 34
  Week 4: Suicidal thoughts: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Suicidal thoughts | 10 | 3 | 10
  Week 4: Suicidal thoughts w/ method: number analyzed (Participants) | 11 | 3 | 12
  Week 4: Suicidal thoughts w/ method | 4 | 0 | 5
  Week 4: Suicidal intent (w/o plan): number analyzed (Participants) | 11 | 3 | 12
  Week 4: Suicidal intent (w/o plan) | 1 | 0 | 1
  Week 4: Suicidal intent w/ plan: number analyzed (Participants) | 11 | 3 | 12
  Week 4: Suicidal intent w/ plan | 1 | 0 | 0
  Week 8: Wish to be dead: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Wish to be dead | 19 | 6 | 15
  Week 8: Suicidal thoughts: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Suicidal thoughts | 6 | 2 | 2
  Week 8: Suicidal thoughts w/ method: number analyzed (Participants) | 6 | 2 | 2
  Week 8: Suicidal thoughts w/ method | 3 | 0 | 0
  Week 8: Suicidal intent (w/o plan): number analyzed (Participants) | 6 | 2 | 2
  Week 8: Suicidal intent (w/o plan) | 0 | 0 | 0
  Week 8: Suicidal intent w/ plan: number analyzed (Participants) | 6 | 2 | 2
  Week 8: Suicidal intent w/ plan | 0 | 0 | 0
  End of Period I: Wish to be dead | 32 | 8 | 26
  End of Period I: Suicidal thoughts | 13 | 3 | 9
  Endf of Period I: Suicidal thoughts w/ method: number analyzed (Participants) | 16 | 3 | 16
  Endf of Period I: Suicidal thoughts w/ method | 7 | 0 | 7
  End of Period I: Suicidal intent (w/o plan): number analyzed (Participants) | 16 | 3 | 16
  End of Period I: Suicidal intent (w/o plan) | 2 | 0 | 1
  End of Period I: Suicidal intent w/ plan: number analyzed (Participants) | 16 | 3 | 16
  End of Period I: Suicidal intent w/ plan | 1 | 0 | 0

33. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Ideation - Wish to be Dead (Combined Treatment Period I and II)
Description: The C-SSRS is a scale for assessing risk for suicidal behavior and suicide ideation and was administered by the clinician. Affirmative or negative responses were provided to 5 items for suicide ideation (1. Wish to be dead; 2. Suicidal thoughts; 3. Suicidal thoughts with a method (no specific plan or intent to act); 4. Suicidal intent (without a specific plan); 5. Suicidal intent with specific plan. If participants responded with a negative response for questions 1 and 2, the remaining questions are skipped. If question 2 was responded to with a positive response, the remaining questions need to be asked. Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-10.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 (Placebo/FK949E only from week 12, FK949E 150 mg/FK949E & FK949E 300 mg/FK949E from week 4)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 14 | 34
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 6 | 15
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 17 | 9 | 21
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 9 | 8 | 22
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 6 | 8 | 12
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 5 | 5 | 8
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 4 | 4 | 8
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 6 | 4 | 9
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 2 | 4 | 8
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 3 | 4 | 6
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 3 | 3 | 7
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 3 | 4 | 7
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 1 | 4 | 3
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 6 | 11 | 26

34. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Ideation - Suicidal Thoughts (Combined Treatment Period I and II)
Description: as for outcome 33
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Number; unit: particpants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
particpants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 3 | 10
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 2 | 2
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 4 | 2 | 1
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 2 | 2 | 5
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 2 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 1 | 2
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 1 | 2
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 1 | 2
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 2 | 1
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 2
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 1 | 2
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 1 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 2 | 2 | 14

35. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Ideation - Suicidal Thoughts With Method (Combined Treatment Period I and II)
Description: as for outcome 33
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 3 | 12
  Week 4 |  | 0 | 5
  Week 8: number analyzed (Participants) | 0 | 2 | 3
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 4 | 2 | 1
  Week 12 | 1 | 0 | 0
  Week 16: number analyzed (Participants) | 2 | 2 | 5
  Week 16 | 1 | 0 | 4
  Week 20: number analyzed (Participants) | 0 | 2 | 0
  Week 20 |  | 0 |
  Week 24: number analyzed (Participants) | 0 | 2 | 2
  Week 24 |  | 0 | 2
  Week 28: number analyzed (Participants) | 0 | 1 | 2
  Week 28 |  | 0 | 0
  Week 32: number analyzed (Participants) | 1 | 0 | 0
  Week 32 | 1 |  |
  Week 36: number analyzed (Participants) | 0 | 1 | 2
  Week 36 |  | 0 | 2
  Week 40: number analyzed (Participants) | 0 | 2 | 1
  Week 40 |  | 2 | 0
  Week 44: number analyzed (Participants) | 0 | 0 | 2
  Week 44 |  |  | 0
  Week 48: number analyzed (Participants) | 0 | 1 | 2
  Week 48 |  | 1 | 0
  Week 52: number analyzed (Participants) | 0 | 1 | 0
  Week 52 |  | 1 |
  End of combined treatment period: number analyzed (Participants) | 4 | 8 | 27
  End of combined treatment period | 2 | 4 | 12

36. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Ideation - Suicidal Intent Without a Plan (Combined Treatment Period I and II)
Description: as for outcome 33
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 3 | 12
  Week 4 |  | 0 | 1
  Week 8: number analyzed (Participants) | 0 | 2 | 3
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 4 | 2 | 1
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 2 | 2 | 5
  Week 16 | 1 | 0 | 1
  Week 20: number analyzed (Participants) | 0 | 2 | 0
  Week 20 |  | 0 |
  Week 24: number analyzed (Participants) | 0 | 2 | 2
  Week 24 |  | 0 | 2
  Week 28: number analyzed (Participants) | 0 | 1 | 2
  Week 28 |  | 0 | 0
  Week 32: number analyzed (Participants) | 1 | 0 | 0
  Week 32 | 1 |  |
  Week 36: number analyzed (Participants) | 0 | 1 | 2
  Week 36 |  | 0 | 0
  Week 40: number analyzed (Participants) | 0 | 2 | 1
  Week 40 |  | 0 | 0
  Week 44: number analyzed (Participants) | 0 | 0 | 2
  Week 44 |  |  | 0
  Week 48: number analyzed (Participants) | 0 | 1 | 2
  Week 48 |  | 1 | 0
  Week 52: number analyzed (Participants) | 0 | 1 | 0
  Week 52 |  | 0 |
  End of combined treatment period: number analyzed (Participants) | 4 | 8 | 27
  End of combined treatment period | 2 | 1 | 4

37. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Ideation - Suicidal Intent With a Plan (Combined Treatment Period I and II)
Description: as for outcome 33
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 3 | 12
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 2 | 3
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 4 | 2 | 1
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 2 | 2 | 5
  Week 16 | 1 | 0 | 0
  Week 20: number analyzed (Participants) | 0 | 2 | 0
  Week 20 |  | 0 |
  Week 24: number analyzed (Participants) | 0 | 2 | 2
  Week 24 |  | 0 | 0
  Week 28: number analyzed (Participants) | 0 | 1 | 2
  Week 28 |  | 0 | 0
  Week 32: number analyzed (Participants) | 1 | 0 | 0
  Week 32 | 1 |  |
  Week 36: number analyzed (Participants) | 0 | 1 | 2
  Week 36 |  | 0 | 0
  Week 40: number analyzed (Participants) | 0 | 2 | 1
  Week 40 |  | 0 | 0
  Week 44: number analyzed (Participants) | 0 | 0 | 2
  Week 44 |  |  | 0
  Week 48: number analyzed (Participants) | 0 | 1 | 2
  Week 48 |  | 0 | 0
  Week 52: number analyzed (Participants) | 0 | 1 | 0
  Week 52 |  | 0 |
  End of combined treatment period: number analyzed (Participants) | 4 | 8 | 27
  End of combined treatment period | 2 | 0 | 1

38. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors (Treatment Period I)
Description: The C-SSRS is a scale for assessing risk for suicidal behavior and suicide ideation and was administered by the clinician. Affirmative or negative responses were provided to 7 items to suicidal behaviors (1. suicide attempt; 2. Self-injury without suicide intent; 3. discontinued suicide attempt; 4. interrupted suicide attempt; 5. preliminary action to suicide; 6. suicidal behavior; 7. completed suicide).
Time Frame: Weeks 4, 8
Population: SAF participants with available data at each time point; LOCF imputation method was used for end of Treatment Period I.
Measure: Number; unit: participants
Arm/Group | Placebo | FK949E 150 mg | FK949E 300 mg
Number analyzed (Participants) | 173 | 73 | 176
participants
  Week 4: Suicide attempt: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Suicide attempt | 0 | 0 | 0
  Week 4: Self-injury w/o intent: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Self-injury w/o intent | 1 | 0 | 2
  Week 4: Discontinued attempt: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Discontinued attempt | 0 | 0 | 0
  Week 4: Interrupted attempt: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Interrupted attempt | 0 | 0 | 0
  Week 4: Preliminary act to suicide: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Preliminary act to suicide | 0 | 0 | 0
  Week 4: Suicidal behavior: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Suicidal behavior | 0 | 0 | 0
  Week 4: Completed suicide: number analyzed (Participants) | 160 | 68 | 159
  Week 4: Completed suicide | 0 | 0 | 0
  Week 8: Suicide attempt: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Suicide attempt | 0 | 0 | 0
  Week 8: Self-injury w/o intent: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Self-injury w/o intent | 0 | 0 | 2
  Week 8: Discontinued attempt: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Discontinued attempt | 0 | 0 | 0
  Week 8: Interrupted attempt: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Interrupted attempt | 0 | 0 | 0
  Week 8: Preliminary act to suicide: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Preliminary act to suicide | 0 | 0 | 0
  Week 8: Suicidal behavior: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Suicidal behavior | 0 | 0 | 0
  Week 8: Completed suicide: number analyzed (Participants) | 136 | 60 | 140
  Week 8: Completed suicide | 0 | 0 | 0
  End of Period I: Suicide attempt | 2 | 0 | 0
  End of Period I: Self-injury w/o intent | 1 | 0 | 2
  End of Period I: Discontinued attempt | 0 | 0 | 0
  End of Period I: Interrupted attempt | 0 | 0 | 0
  End of Period I: Preliminary act to suicide | 0 | 0 | 0
  End of Period I: Suicidal behavior | 2 | 0 | 0
  End of Period I: Completed suicide | 0 | 0 | 0

39. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Suicide Attempt (Combined Treatment Period I and II)
Description: The C-SSRS is a scale for assessing risk for suicidal behavior and suicide ideation and was administered by the clinician. Affirmative or negative responses were provided to 7 items to suicidal behaviors (1. suicide attempt; 2. Self-injury without suicide intent; 3. discontinued suicide attempt; 4. interrupted suicide attempt; 5. preliminary action to suicide; 6. suicidal behavior; 7. completed suicide). Baseline for Placebo / FK949E was at week 12 therefore no data were calculated for weeks 1-10.
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 1
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 1 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 0
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 1 | 1 | 1

40. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Self-injury Behavior Without Intent (Combined Treatment Period I and II)
Description: as for outcome 39
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 2
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 2
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 1
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 1 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 1 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 1
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 1
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 0 | 1
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 0 | 0 | 1

41. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Discontinued Attempt (Combined Treatment Period I and II)
Description: as for outcome 39
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 0
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 1 | 0
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  Endof combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  Endof combined treatment period | 0 | 0 | 0

42. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Interrupted Attempt (Combined Treatment Period I and II)
Description: as for outcome 39
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 0
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 1 | 0 | 0

43. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Preliminary Act to Suicide (Combined Treatment Period I and II
Description: as for outcome 39
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 0
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Suicidal Behavior (Combined Treatment Period I and II)
Description: as for outcome 39
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 1
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 1 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 0
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 1 | 0
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 2 | 1 | 1

45. Secondary Outcome: Number of Participants With an Affirmative Response to C-SSRS: Suicidal Behaviors - Completed Suicide (Combined Treatment Period I and II)
Description: as for outcome 39
Time Frame: as for outcome 33
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo / FK949E | FK949E 150 mg / FK949E | FK949E 300 mg / FK949E
Number analyzed (Participants) | 120 | 74 | 179
Participants
  Week 4: number analyzed (Participants) | 0 | 68 | 159
  Week 4 |  | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 60 | 140
  Week 8 |  | 0 | 0
  Week 12: number analyzed (Participants) | 120 | 51 | 123
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 112 | 49 | 118
  Week 16 | 0 | 0 | 0
  Week 20: number analyzed (Participants) | 103 | 47 | 115
  Week 20 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 101 | 42 | 111
  Week 24 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 96 | 38 | 105
  Week 28 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 89 | 36 | 98
  Week 32 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 85 | 35 | 92
  Week 36 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 83 | 33 | 88
  Week 40 | 0 | 0 | 0
  Week 44: number analyzed (Participants) | 81 | 33 | 83
  Week 44 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 81 | 32 | 76
  Week 48 | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 79 | 32 | 74
  Week 52 | 0 | 0 | 0
  End of combined treatment period: number analyzed (Participants) | 120 | 73 | 176
  End of combined treatment period | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Groups:
- Treatment Period I: Placebo: Participants received placebo administered orally once daily at bedtime for 8 weeks in Treatment Period I. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
- Treatment Period I: FK949E 150 mg: After 2 days of up-titration, participants received FK949E 150 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
- Treatment Period I: FK949E 300 mg: After 4 days of up-titration, participants received FK949E 300 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. If transition criteria were not met, participants underwent to a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
- Treatment Period I + II: Placebo / FK949E: Participants received placebo administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive placebo for 4 weeks, followed by a 1-week dose adjustment period, and a treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
- Treatment Period I + II: FK949E 150 mg / FK949E: Participants received FK949E 150 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive FK949E 150 mg for 4 weeks followed by a 1-week dose-adjustment period and a treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
- Treatment Period I + II: FK949E 300 mg / FK949E: Participants received FK949E 300 mg administered orally once daily at bedtime for 8 weeks in Treatment Period I. Participants who met the transition criteria continued to Treatment Period II which consisted of a transition period in which participants continued to receive FK949E 300 mg for 4 weeks followed by a 1-week dose-adjustment period and a treatment period in which participants received either open-label FK949E 150 mg or 300 mg (depending on dose increase or reduction guidelines) administered orally for 39 weeks. Participants underwent a dose-tapering period (1 week) and a follow-up period (1 week) thereafter.
Arm/Group | Treatment Period I: Placebo | Treatment Period I: FK949E 150 mg | Treatment Period I: FK949E 300 mg | Treatment Period I + II: Placebo / FK949E | Treatment Period I + II: FK949E 150 mg / FK949E | Treatment Period I + II: FK949E 300 mg / FK949E
All-Cause Mortality (participants affected / at risk) | 2/177 | 0/74 | 0/179 | 0/120 | 0/74 | 0/179
Serious Adverse Events (participants affected / at risk) | 2/177 | 1/74 | 0/179 | 1/120 | 4/74 | 5/179
Other Adverse Events (participants affected / at risk) | 62/177 | 51/74 | 140/179 | 106/120 | 59/74 | 164/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period I: Placebo (N=177) | Treatment Period I: FK949E 150 mg (N=74) | Treatment Period I: FK949E 300 mg (N=179) | Treatment Period I + II: Placebo / FK949E (N=120) | Treatment Period I + II: FK949E 150 mg / FK949E (N=74) | Treatment Period I + II: FK949E 300 mg / FK949E (N=179)
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period I: Placebo (N=177) | Treatment Period I: FK949E 150 mg (N=74) | Treatment Period I: FK949E 300 mg (N=179) | Treatment Period I + II: Placebo / FK949E (N=120) | Treatment Period I + II: FK949E 150 mg / FK949E (N=74) | Treatment Period I + II: FK949E 300 mg / FK949E (N=179)
Palpitation (Cardiac disorders) | 2 | 2 | 0 | 2 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 6 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 1 | 2 | 3 | 1
Hyperprolactinemia (Endocrine disorders) | 1 | 0 | 4 | 2 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2 | 7 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 4 | 7
Constipation (Gastrointestinal disorders) | 3 | 10 | 14 | 6 | 16 | 21
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 4 | 3 | 6 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 3 | 2 | 2 | 5 | 6 | 10
Vomiting (Gastrointestinal disorders) | 4 | 3 | 1 | 0 | 7 | 5
Malaise (General disorders) | 2 | 3 | 16 | 12 | 6 | 22
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 2 | 2
Thirst (General disorders) | 5 | 9 | 50 | 17 | 12 | 51
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 4
Cystitis (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 3 | 1 | 9
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 4 | 2
Nasopharyngitis (Infections and infestations) | 19 | 12 | 26 | 40 | 36 | 58
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 2 | 2 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 1 | 5
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | 1
Wound (Injury, poisoning and procedural complications) | 4 | 0 | 3 | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 0 | 4 | 8 | 2 | 5 | 13
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 2 | 3 | 5 | 5
Blood creatinine phosphokinase increased (Investigations) | 1 | 7 | 5 | 8 | 9 | 13
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0
Blood prolactin increased (Investigations) | 5 | 4 | 13 | 5 | 6 | 21
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 3 | 2
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 3 | 1 | 1 | 5
Blood triglycerides increased (Investigations) | 2 | 3 | 3 | 3 | 6 | 9
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 3 | 3 | 3 | 4
Weight increased (Investigations) | 0 | 1 | 8 | 19 | 5 | 19
Tri-iodothyronine free increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 13 | 2 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 6 | 2 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 1 | 5
Akathisia (Nervous system disorders) | 4 | 7 | 15 | 9 | 9 | 21
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Bradykinesia (Nervous system disorders) | 0 | 0 | 2 | 3 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 4 | 5 | 3 | 9 | 7
Dizziness postural (Nervous system disorders) | 2 | 0 | 7 | 3 | 0 | 9
Dystonia (Nervous system disorders) | 0 | 0 | 1 | 4 | 0 | 3
Headache (Nervous system disorders) | 2 | 1 | 3 | 7 | 5 | 12
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 3 | 0 | 4
Somnolence (Nervous system disorders) | 4 | 26 | 80 | 59 | 34 | 97
Depression (Psychiatric disorders) | 10 | 1 | 4 | 2 | 5 | 8
Hypomania (Psychiatric disorders) | 4 | 0 | 1 | 1 | 0 | 5
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 5 | 2 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment.